CLINICAL TRIAL: NCT02014935
Title: Immediate Effect of Low Intensity Laser on the Spastic Muscle Fatigued.
Brief Title: Immediate Effect of Laser on Spasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratório de Engenharia de Reabilitação Sensorio Motora (Other)
Responsible Party: Principal Investigator, Djenifer Queiroz de Souza, Mariana César Ribeiro dos Reis, Laboratório de Engenharia de Reabilitação Sensorio Motora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 1542193200005503
Record Dates: First submitted 2013-11-07; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Ischemic Brain
Keywords: Low-intensity Laser; Spasticity; pain,; Fatigue
MeSH Terms: conditions — Muscle Spasticity; Pain; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low intensity laser (Experimental): So that this research recrutarou 30 subjects with spastic hemiparesis sequel, post stroke who have gone through three phases, with three evaluations. If this conformation is necessary, therefore, it is a search for intergroup analysis, and the values found in Phase I were faced with the values found in Phases II and III.
  The phases comprise:
  * Phase I (1st Cycle): Individuals treated with LLLT not only performed the evaluation of muscle activity, torque and lactic acid level.
  * Phase II (2nd Cycle): Individuals undergoing the application of LLLT, with the same off, and assessment of muscle activity, torque and lactic acid level.
  * Phase III (3rd Cycle): Individuals undergoing the application of LILT and evaluation of muscle activity, torque and lactic acid level.
  Interventions: Other: Low intensity laser

INTERVENTIONS:
Other: Low intensity laser — The study wants to evaluate the use of low intensity laser on the spastic muscle.
  Want to assess whether the Low level laser prove change in muscle performace of the individual but also alters muscle activity and blood lactate.

SUMMARY:
The poor eating habits and sedentary lifestyle of young people can reflect on structural changes in adult life, leading to vascular brain diseases. The cerebrovascular accident (AVC) represents the second cause of death throughout the country. Presents rapid development of clinical signs, providing focal disorders or brain function. It is necessary to the knowledge and development of new treatment techniques that may minimize the sequelae caused by the AVC, which is a common disease and of great impact on public health, represents the main cause of adult neurological disability, affecting the basic functions of the limbs, motor control and balance, strength and mobility, which involves changes in daily life and low self-esteemIn addition to the high cost of treatment and in the long run.

Thus, this study aims to analyze the response of low intensity laser on the prevention of pain and fatigue induced in rectus femoris, vastus of patients with sequelae of spasticity associated with effects on the laser promotes on muscle performance and muscle activity.

It is believed that this study get positive results as regards the increase of time antecedent to muscular fatigue associated with the skeletal muscle performance, so that the normotonics muscles gain strength and overcome the resistance of hypertonic muscles. In this way, it is expected that after the application of low intensity Laser Therapy (LILT) occurs to the adequacy of spasticity, muscle function the gain that had provided the highest quality of physiotherapy care.

It is known that treatment with the laser on the skeletal musculature, presents positive results and on the peak torque, by means of the skeletal muscle performance and consequently gain increase muscle performance (LEAL JUNIOR et al, 2010; ALMEIDA et al, 2011).

Armed with this information you can infer that the low intensity laser therapy on the spastic muscle, would result in improving muscle performance, with an increase of pre-stressing, improving the functional capacity of individuals under the exercises imposed by physical therapy. In this way, the sessions will take more satisfactory results which jointly provided better quality of life for these patients.

DETAILED DESCRIPTION:
With the course of the years, became notorious the transformation in the epidemiological profile of the Brazilian population, with the progressive decline of infectious diseases and illness narratives and the gradual growth of the chronic degenerative diseases, particularly cardiovascular diseases of (ARAÚJO, 2012)

According to statistics of the Ministry of health, in the year 2010 were recorded about 100 thousand deaths due to cerebrovascular accident (AVE), a result of the sudden interruption of blood flow of the brain, which is currently responsible for leading cause death in Brazil (MINISTRY of health, 2012).

The heterogeneity of the Brazilian population, would explain the current epidemiological transition, and as a result the high rates of mortality. The diseases of the circulatory system are as main cause death of Brazil, emphasizing the cerebrovascular disease, responsible for one third of deaths in the country.

The cerebral arteries are responsible for giving the necessary nutrients as a source of energy to neurons, the brain requires intense blood flow to meet your high intake of nutrients. Being that the interruption of the flow of oxygen and glucose for a period in excess of five minutes can cause irreversible damage to the brain.

Several pathological processes can cause the interruption of blood flow in certain brain areas. Between these processes include hemorrhages, embolisms, stroke and diseases that lead to suspension of blood flow, and therefore the deficit in the supply of nutrients.

The blood deficit promotes changes in cellular metabolism, which can lead to injury and/or death of brain tissue. According to estimates, 80% of the incidence of BIRD arteriolar occlusion resulting from atheroma plates or secondary brain artery emboli that deprive the brain of blood supply.

The likelihood of the AVE doubles every decade of life, from 55 years of age. Although leverage the ranking of deaths in the country, statistics from the Ministry of health in 2010, showed decreased mortality rate in the age group up to 70 years, representing an annual average reduction of 3.2% (MINISTRY of health, 2012).

As established earlier, the differences in the prevalence of risk factors among the population due to high heterogeneity, that is, different customs, habits and lifestyles. So in that, poor eating habits and physical youth population may reflect structural changes in adulthood, and may lead to vascular brain diseases. Among the risk factors associated with the AVE is hypertension, dyslipidemias, diabetes, smoking, alcoholism.

In general the clinical picture presents itself with motor and sensory changes, that may be associated with deficits in cognitive and perceptual functions by damaging both physical and physiological functions of the patient (DIETZ; SINKJAER, 2007). Due to the AVE be associated with motor disability tables, resulting in physical limitations, mainly resulting from spasticity, is necessary to search for ways to minimise this damage. In this way, it is believed that with the help of biomedical instrumentation, which in addition to providing quantitative and reliable data on the functional capacity of the individual, allows the development and recruitment of equipment to help in the evaluation of the General State of the patient and so consequently best results before the practice of neurological rehabilitation. Therefore it is of utmost importance to biomedical resource utilization as surface electromyography that refers to a method of non-invasive monitoring, providing values for the square root of the mean squared Value (RMS - R Englishoot Mean Square), demonstrating this parameter the results of signal amplitude through the average power in the time interval analyzed, containing information about the amount of traction units fired at any given movement

Isokinetic dynamometry bound that provides resistance to joint movement over a given range, enabling the analysis of muscle force-related parameters such as torque, power, and endurance. These two features combined will contribute to the determination of the time when the o muscle spastics had to fatigue muscles. On this information, the sessions can be reworded to the concrete limitations of patients and consequently the improvement of rehabilitation, which will automatically improves the quality of life of these individuals.

ELIGIBILITY:
Inclusion Criteria:

* People with spastic hemiparesis;

  * Medical referral for physiotherapy;
  * Age between 40 and 80 years;
  * Women who are in menopause;
  * Cognitive preserved, being able to respond to verbal stimuli;
  * Modified Ashworth scale, with a maximum of 2 degree of spasticity in the flexor muscles of the knee, specifically in the muscles that make up the Quadriceps femoris.

Exclusion Criteria:

* · Patients with Hypoesthesia and/or Hyperesthesia of the side to be studied

  * The presence of active infection and rashes at the site of application of the electrodes;
  * Joint stiffness, contractures and deformities;
  * Broca's aphasia
  * Uncontrolled arterial hypertension;
  * Presence of neoplastic lesion at the site of application;
  * Intake of analgesics and/or anti-inflammatory medication during the two weeks of evaluation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
muscle activity | three days
  Muscle activity will be captured with the aid of electromyography. So that the EMG data will be collected with the completion of the isometric contraction of the rectus femoris, vastus. Being held in this capture period of 50 seconds.

SECONDARY OUTCOMES:
muscular performance | three days
  The muscular performance will be analyzed with the equipment isokinetic dynamometer.
  Volunteers will be placed in a sitting position in the chair equipment (Biodex System ®), with the limb to be assessed on the supported equipment support.
  Thus the device is triggered mode isometric contraction and the individual remained in contraction for a time of 50 seconds. Patients will be advised to carry their maximum contraction so as to obtain the torque of the muscles.

OTHER OUTCOMES:
blood lactate | three days
  The collection of blood lactate happen with the aid of lactomer , portable device brand (Accutrend ® PLUS Roche). Will be collected before and after the completion of the exercise isometric contraction, a drop of blood to detect the level of lactate in the blood. So to differentiate the amount found in the blood before and after exercise and to see whether the application of Laser alter this concentration in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana C Reis, Therapy, Principal Investigator — University of Vale do Paraiba
Locations (1):
- Universidade do Vale do Paraíba, São José dos Campos, São Paulo, Brazil

REFERENCES:
- [Background] ALMEIDA, P., et al. Red (660nm) and infrared (830nm) low-level laser therapy in skeletal muscle fatigue in humans: what is better?. Lasers in a Medical Science., v.27, p.453-458, 2012. LEAL JUNIOR, E. C., et al. Effects of low level laser therapy (LLLT) in the development of exercise-induced skeletal muscle fatigue and changes in biochemical markers related to post- exercise recovery. Journal of Orthopaedic & Sports Physical Therapy., v.40, n.8, p.524-32, 2010. DIETZ, V.; SINKJAER, T. Spastic movement disorder:impaired reflex function and altered muscle mechanics Review. Lancet Neurology., v.6, p.725-733, 2007. MINISTÉRIO DA SAÚDE SÃO PAULO: banco de dados. Disponível em: http://portalsaude.saude.gov.br/portalsaude/noticia/7904/162/avc:-governo-alerta-para-%3Cbr%3Eprincipal-causa-de-mortes.html. STROKE, 2006. In:World Health Organization. Neurological disordes: public health challenges. Geneva: World Health Organization, 2006. p.163-175.
- See also: This study serves as a reference of the protocol being carried out. — http://www.ncbi.nlm.nih.gov/pubmed/19057981